CLINICAL TRIAL: NCT05755997
Title: A Randomized, Double-blind, Single-centre, Two-period Cross-over, Placebo-controlled Trial on Safety and Efficacy in Patients With Genetically Proven CADASIL
Brief Title: CERebrolysin In CADASIL
Acronym: CERICA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ever Neuro Pharma GmbH (Industry)
Collaborators: idv Datenanalyse & Versuchsplanung (Unknown); XClinical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVER-CZ-0421; 2022-002394-29 (EudraCT Number)
Record Dates: First submitted 2023-02-14; First posted 2023-03-06 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cadasil
MeSH Terms: conditions — CADASIL | interventions — cerebrolysin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A two-period cross-over design, in which participants will be randomly allocated to either the Verum-Control sequence (sequence 1) or the Control-Verum sequence (sequence 2) in a 1:1 randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group 1 (Other): Cerebrolysin - Placebo
  Interventions: Drug: Cerebrolysin; Drug: 0.9 % NaCl
- Study group 2 (Other): Placebo - Cerebrolysin
  Interventions: Drug: Cerebrolysin; Drug: 0.9 % NaCl

INTERVENTIONS:
Drug: Cerebrolysin — 40 ml Cerebrolysin and 60 ml 0.9% NaCl per day for 4 days every month for 1 year
  Other Names: Renacenz
Drug: 0.9 % NaCl — 100 ml 0.9% NaCl per day for 4 days every month for 1 year
  Other Names: Sodium Chloride

SUMMARY:
The objective of this trial is the global risk-benefit assessment of Cerebrolysin as compared to Placebo in patients with genetically proven CADASIL. In addition, a traditional approach will be taken based on an evaluation of the separate risk and benefit domains in comparison with placebo.

DETAILED DESCRIPTION:
Safety data area collected throughout the study (adverse events, vital signs and laboratory tests) and thereafter in case of ongoing serious adverse events (SAEs) at study endpoint.

Optional secondary parameters include analyses of biomarkers (samples of blood, hair, urine, and saliva).

ELIGIBILITY:
Inclusion Criteria:

1. Patients of ≥18 years of age, all genders
2. Diagnosis of CADASIL based on clinical symptoms, MRI, and genetic analysis
3. MoCA >11
4. Adequate visual, auditory, and language skills (no language interpreter required) to follow study procedures
5. Patient is not of childbearing potential (i.e. women are post-menopausal for two years, surgically sterile, or using adequate method of contraception)
6. Patient participates voluntarily and gave written informed consent

Exclusion Criteria:

1. Any significant neurological disease/conditions other than CADASIL
2. Focal lesions that may be responsible for the cognitive status of the patient (e.g.

   infectious disease, space-occupying lesion, normal pressure hydrocephalus)
3. Any other diseases/conditions that may affect compliance with the protocol, such as:

   1. severe psychiatric disorders within the last three months
   2. delusional symptoms
   3. history of schizophrenia, schizoaffective disorder, bipolar affective disorder
   4. major depressive disorder newly identified within eight weeks before screening
   5. history of alcohol or substance abuse or dependence within the past two years
4. Any circumstances that -in the investigator's opinion- may result in the patient's non-compliance with study procedures, e.g. fragile or thin veins that prevent many i.v. infusions
5. Any other disease/conditions that may affect the safety assessment, such as:

   1. history of systemic cancer within the past two years
   2. history of myocardial infarction in the past year or unstable or severe cardiovascular disease (including uncontrolled hypertension and/or history of unstable hypertension not compensated by antihypertensive therapy)
   3. any clinically significant laboratory abnormalities at screening
   4. uncontrolled insulin-requiring diabetes or non-insulin dependent diabetes mellitus (HbA1c >87 mmol/mol)
6. Use of concomitant medication with neuroprotective/neurotrophic/nootropic effects (e.g. ginkgo biloba, erythropoietin, citicoline, amantadine, piracetam)
7. Any condition that would represent a contraindication for Cerebrolysin administration:

   1. hypersensitivity to one of the components of the drug
   2. epilepsy
   3. severe renal impairment (estimated Glomerular Filtration Rate [eGFR] <30 ml/min/1.73 m2 as assessed at local laboratory within one month before screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive battery (RAVLT) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Rey Auditory Verbal Learning Test (AVLT)
Change in cognitive battery (ROCF: Copy, immediate recall) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Rey-Osterrieth Complex Figure Test (ROCF): Copy, immediate recall
Change in cognitive battery (Digit Symbol Coding, subscale of WAIS-PSI) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Digit Symbol Coding (subscale of WAIS-PSI)
Change in cognitive battery (Digit Span: Digit backward (subscale of WAIS-WMI) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Digit Span: Digit backward (subscale of WAIS-WMI)
Change in cognitive battery (Trail Making Test, Part B) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Trail Making Test (Part B)
Change in cognitive battery (ROCF: Delayed recall) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Rey-Osterrieth Complex Figure Test (ROCF): Delayed recall
Change in cognitive battery (Stroop Color and Word Test - Prague Version) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Stroop Color and Word Test - Prague Version (word/dots interference)
Change in cognitive battery (MoCA) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Montreal Cognitive Assessment (MoCA)
Change in mood (Beck Depression Inventory-II) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Beck Depression Inventory-II (BDI-II)
Change in imaging (White matter lesion volume) | Baseline, Month 12, Month 27
  - White matter lesion volume (MRI)

SECONDARY OUTCOMES:
Change in cognitive battery, secondary outcome (Spatial Pattern Separation Task) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Spatial Pattern Separation Task
Change in cognitive battery, secondary outcome (Navigation Test Suite) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Navigation Test Suite
Change in cognitive battery, secondary outcome (Trail Making Test, Part A) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Trail Making Test (Part A)
Change in cognitive battery, secondary outcome (Stroop Color and Word Test - Prague Version) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Stroop Color and Word Test - Prague Version (color-word/dots interference)
Change in cognitive battery, secondary outcome (Symbol Search, subscale of WAIS-PSI) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Symbol Search (subscale of WAIS-PSI)
Change in cognitive battery, secondary outcome (Digit Span: Digit forward, subscale of WAIS-WMI) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Digit Span: Digit forward (subscale of WAIS-WMI)
Change in mood, secondary outcome (Beck Anxiety Inventory) | Baseline, Month 6, Month 12, Month 21, Month 27
  - Beck Anxiety Inventory
Change in neurological deficits, secondary outcome (NIH stroke scale) | Baseline, Month 6, Month 12, Month 21, Month 27
  - NIH stroke scale (NIHSS)
Change in imaging, secondary outcome (Index of general cortical thinning) | Baseline, Month 12, Month 27
  - Index of general cortical thinning (MRI)
Change in imaging, secondary outcome (Post-stroke lacune volume) | Baseline, Month 12, Month 27
  - Post-stroke lacune volume (MRI)
Change in biomarker analysis, secondary outcome (Neurofilament light chain) | Baseline, Month 12, Month 27
  - Neurofilament light chain (NFL)

OTHER OUTCOMES:
Experimental (to be defined after study endpoint): Change in Serotonin level (hair, mean) | Baseline, Month 12, Month 27
  - mean over several weeks
Experimental (to be defined after study endpoint): Change in Oxytocin level (hair, mean) | Baseline, Month 12, Month 27
  - mean over several weeks
Experimental (to be defined after study endpoint): Change in Cortisol level (hair, mean) | Baseline, Month 12, Month 27
  - mean over several weeks
Experimental (to be defined after study endpoint): Change in Serotonin level (hair, greyish level) | Baseline, Month 12, Month 27
  - hair color (greyish level)
Experimental (to be defined after study endpoint): Change in Oxytocin level (hair, greyish level) | Baseline, Month 12, Month 27
  - hair color (greyish level)
Experimental (to be defined after study endpoint): Change in Cortisol level (hair, greyish level) | Baseline, Month 12, Month 27
  - hair color (greyish level)
Experimental (to be defined after study endpoint): Change in Serotonin level (saliva, day value) | Baseline, Month 12, Month 27
  - value of this time at this day
Experimental (to be defined after study endpoint): Change in Oxytocin level (saliva, day value) | Baseline, Month 12, Month 27
  - value of this time at this day
Experimental (to be defined after study endpoint): Change in Cortisol level (saliva, day value) | Baseline, Month 12, Month 27
  - value of this time at this day
Experimental (to be defined after study endpoint): Change in Serotonin level (saliva, epigenetic age) | Baseline, Month 12, Month 27
  - epigenetic age
Experimental (to be defined after study endpoint): Change in Oxytocin level (saliva, epigenetic age) | Baseline, Month 12, Month 27
  - epigenetic age
Experimental (to be defined after study endpoint): Change in Cortisol level (saliva, epigenetic age) | Baseline, Month 12, Month 27
  - epigenetic age
Experimental (to be defined after study endpoint): Change in Serotonin level (blood pellet, epigenetic age) | Baseline, Month 12, Month 27
  - epigenetic age
Experimental (to be defined after study endpoint): Change in Oxytocin level (blood pellet, epigenetic age) | Baseline, Month 12, Month 27
  - epigenetic age
Experimental (to be defined after study endpoint): Change in Cortisol level (blood pellet, epigenetic age) | Baseline, Month 12, Month 27
  - epigenetic age
Experimental (to be defined after study endpoint): Change in Serotonin level (blood pellet, omega-3 fatty acids) | Baseline, Month 12, Month 27
  - omega-3 fatty acids
Experimental (to be defined after study endpoint): Change in Oxytocin level (blood pellet, omega-3 fatty acids) | Baseline, Month 12, Month 27
  - omega-3 fatty acids
Experimental (to be defined after study endpoint): Change in Cortisol level (blood pellet, omega-3 fatty acids) | Baseline, Month 12, Month 27
  - omega-3 fatty acids
Experimental (to be defined after study endpoint): Change in Serotonin level (blood plasma) | Baseline, Month 12, Month 27
  - somascan
Experimental (to be defined after study endpoint): Change in Oxytocin level (blood plasma) | Baseline, Month 12, Month 27
  - somascan
Experimental (to be defined after study endpoint): Change in Cortisol level (blood plasma) | Baseline, Month 12, Month 27
  - somascan
Experimental (to be defined after study endpoint): Change in Serotonin level (urine, alpha klotho) | Baseline, Month 12, Month 27
  - alpha klotho
Experimental (to be defined after study endpoint): Change in Oxytocin level (urine, alpha klotho) | Baseline, Month 12, Month 27
  - alpha klotho
Experimental (to be defined after study endpoint): Change in Cortisol level (urine, alpha klotho) | Baseline, Month 12, Month 27
  - alpha klotho
Experimental (to be defined after study endpoint): Change in Serotonin level (urine, epigenetic markers) | Baseline, Month 12, Month 27
  - epigenetic markers
Experimental (to be defined after study endpoint): Change in Oxytocin level (urine, epigenetic markers) | Baseline, Month 12, Month 27
  - epigenetic markers
Experimental (to be defined after study endpoint): Change in Cortisol level (urine, epigenetic markers) | Baseline, Month 12, Month 27
  - epigenetic markers
Experimental (to be defined after study endpoint): Change in capillary permeability (Ktrans) in grey and white matter | Baseline, Month 12, Month 27
  Capillary permeability (Ktrans) in grey and white matter (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Aleš Tomek, MUDr., Ph.D., Principal Investigator — Motol University Hospital
Locations (1):
- Motol University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No